CLINICAL TRIAL: NCT02521142
Title: Non-invasive Optical Angiography in Age-related Macular Degeneration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Prof. Dr., Medical University of Vienna
Other Study IDs: NOAA
Record Dates: First submitted 2015-08-03; First posted 2015-08-13 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Age Related Macular Degeneration
Keywords: OCT Angiography
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- AMD: treatment-naive
  Interventions: Other: Non-invasive OCT based optical angiography; Other: Oxymap T1; Other: OCT; Other: FLA/ICG angiography
- AMD: active neovascular AMD
  Interventions: Other: Non-invasive OCT based optical angiography; Other: Oxymap T1; Other: OCT; Other: FLA/ICG angiography

INTERVENTIONS:
Other: Non-invasive OCT based optical angiography — This measurement will be obtained after the dilation of the pupil. Optical coherence tomography (OCT) is a non-invasive optical imaging modality enabling cross-sectional tomographic in vivo visualization of internal microstructure in biological systems. In ophthalmology OCT has become a standard device in visualizing the retina and is also considered a standard tool in the diagnosis of retinal disease. In optical angiography blood vessels contrasting against static tissue are visualized in a full depth resolved and label-free manner.
Other: Oxymap T1 — The Oxymap system T1 is installed on a conventional fundus camera (Topcon TRC-50DX), which is operated as for color photography. The Oxymap T1 simultaneously acquires two images of the same area of the fundus at two different wavelengths of light. One of the two wavelengths is sensitive to oxygen saturation, i.e. the light absorbance changes with the oxygen saturation, while the other is insensitive to oxygen saturation and is used to calibrate the light intensity. The two spectral images are automatically processed by the Oxymap Analyzer software. Oxymap Analyzer detects blood vessels and estimates the light absorbance (optical density) at each point along the vessels at each wavelength. The ratio of the optical densities (optical density ratio or ODR) has been shown to be linearly related to hemoglobin oxygen saturation.
Other: OCT — non-invasive imaging of retinal and choroidal structures.
Other: FLA/ICG angiography — Fluorescein Angiography and Indocianine Angiography

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of severe and irreversible visual loss and classified blindness in the elderly throughout Europe and the US. Among these patients, about 6%-8% are afflicted with the advanced stages of AMD, which are responsible for the most severe visual loss. There is now convincing evidence that vascular endothelial growth factor (VEGF) is a major trigger for the formation of pathological choroidal vessels, responsible for the development of the neovascular form of AMD. Today, the gold standard for vascular imaging of the retina and diagnosis of CNV is angiography using fluorescein (FLA) or indocyanine green (ICG), which involves injection of the dye into a vein of the arm. In the recent years tremendous enhancements in the field of optical coherence tomography have been achieved. These developments made it possible to visualize the retinal vasculature in a full depth manner without the application of an intravenous marker. The proposed study tests the hypothesis that visualisation of CNV lesion size with non-invasive OCT angiography is not inferior to FLA/ICG angiography in treatment naïve and previously treated AMD patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients with active CNV due to AMD as assessed by FLA/ICG angiography within 1 week prior to study inclusion

Exclusion criteria

Any of the following will exclude a patient from the study:

* Previous application of intravitreal drugs except anti-VEGF injections
* Active intraocular inflammation
* Presence of an intraocular disease except AMD and cataract

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with CNV due to AMD both, treatment naive and active CNV being treated
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2015-11; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Differences in visualization of lesion size between non-invasive OCT based optical angiography and FLA/ICG angiography in treatment-naïve and treated patients with CNV due to AMD. | Participants will be followed for the duration of outpatient clinic visit, an expected average of 1 days

SECONDARY OUTCOMES:
choroidal thickness as assessed with OCT | participants will be followed for the duration of outpatient clinic visit, an expected average of 1 days
peripapillarly bloodflow as assessed with Doppler OCT | participants will be followed for the duration of outpatient clinic visit, an expected average of 1 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Told R, Reumueller A, Schranz M, Brugger J, Weigert G, Reiter GS, Sacu S, Schmidt-Erfurth U. OCTA Biomarker Search in Patients with nAMD: Influence of Retinal Fluid on Time-Dependent Biomarker Response. Curr Eye Res. 2023 Jun;48(6):600-604. doi: 10.1080/02713683.2023.2184318. Epub 2023 Mar 9. PMID 36891909